CLINICAL TRIAL: NCT01671371
Title: A Randomized, Prospective Study on Point-of-Care Focused Cardiac Ultrasound in Patients Presenting to the Emergency Department With Syncope
Brief Title: Point-of-Care Ultrasound in the Emergency Department Evaluation of Syncope
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to meet enrollment projections
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1110009227
Record Dates: First submitted 2012-07-17; First posted 2012-08-23 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Syncope
Keywords: syncope; point of care; ultrasound; echocardiography
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Ultrasound (Other): A point-of-care ultrasound will be performed during the initial evaluation of the patient after randomization (Defined as Time 0)
  Interventions: Other: Point-of-Care Ultrasound
- Delayed Ultrasound (Other): A point-of-care ultrasound will be performed by the provider at 60 min after initial randomization
  Interventions: Other: Point-of-Care Ultrasound

INTERVENTIONS:
Other: Point-of-Care Ultrasound — Performance of a focused cardiac ultrasound including a qualitative assessment of left ventricular function, pericardial effusion, right ventricular strain, proximal ascending aortic diameter, and inferior vena cava size and collapsibility

SUMMARY:
The purpose of this study is to determine whether point-of-care (bedside) ultrasound assists physicians in the evaluation and management of patients with syncope.

DETAILED DESCRIPTION:
Syncope is one of the more common presentations to the Emergency Department, representing between 1.2-1.5% of all evaluated patients and up to 6% of admissions. Due to an often broad and overlapping differential diagnosis, syncope represents a disease entity that often requires extensive workup. This typically involves laboratory tests, EKGs, x-rays, computed tomography, or other studies that are costly, time-consuming, and, in the case of diagnostic imaging, frequently involves ionizing radiation. Yet, despite extensive testing, an exact diagnosis is not made in up to 50% of cases.

Cardiac causes of syncope include myocardial infarction, pericardial effusion, volume depletion, arrhythmia, among other entities, many of which are life threatening. Echocardiography (cardiac ultrasound) has been used for inpatient syncope evaluations for several decades. In the Emergency Department, echocardiography is currently being used at the point-of-care (POC) in a limited and focused approach to a variety of conditions. However, POC ultrasound has never been systematically evaluated as a diagnostic or prognostic tool specifically for syncope in the Emergency Department. We aim to determine if an ultrasound-based protocol is effective as an adjunct in the evaluation of syncope. Our research study will examine the utility of POC ultrasound in the diagnosis, imaging and laboratory utilization, and prognosis of syncope in the Emergency Department.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older presenting to the ED with acute syncope (defined as transient loss of consciousness) or near syncope (sensation of impending but not actual loss of consciousness) as a reason for ED visit.

Exclusion Criteria:

* persistent altered mental status
* alcohol or illicit drug-related loss of consciousness
* definite seizure, and transient loss of consciousness caused by head trauma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Time to Final Emergency Department Disposition | Time at which an admit or discharge order is placed within the electronic medical record (estimated 2-3 hours)

SECONDARY OUTCOMES:
Time to therapeutic intervention | At onset of therapeutic interventions including but not limited to intravenous fluids and medications (estimated time frame 0 - 6 hours)
Time to clinical procedure | At onset of clinical procedures including but not limited to central line placement, pericardiocentesis, thoracentesis, etc. (estimated time frame 0-6 hours)
Number and Type of other imaging studies | End of Emergency Department Encounter (estimated time frame 1- 6 hours)
  Other imaging studies to included radiographs, additional point-of-care ultrasound, computed tomography, etc.
Information Content provided by Point-of-Care Ultrasound | After performance of point-of-care ultrasound (estimated time frame 1- 6 hours)
  calculating from pre and post test probability estimates and the number of diagnoses
Number and type of laboratory studies | estimated time frame 0-6 hours
Number of and time to consultant services | estimated time frame (0-6 hours)
  Number of consults obtained and the time frame in which the consults were performed

OTHER OUTCOMES:
Short Term Adverse Outcome | 7 days from Emergency Department Visit
  Adverse outcome defined as death, myocardial infarction, arrhythmia, pulmonary embolism, stroke, subarachnoid hemorrhage, significant hemorrhage, or any condition causing a return ED visit and hospitalization for a related event.

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Taylor, M.D., Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Background] Keller C, Tristano JM, De Lorenzo R, et al.
- [Background] Grossman SA, Fischer C, Lipsitz LA, Mottley L, Sands K, Thompson S, Zimetbaum P, Shapiro NI. Predicting adverse outcomes in syncope. J Emerg Med. 2007 Oct;33(3):233-9. doi: 10.1016/j.jemermed.2007.04.001. Epub 2007 Jul 5. PMID 17976548
- [Background] Dhatreecharan S, Azar P, Werner MS, et al.
- [Background] Gabayan GZ, Derose SF, Asch SM, Chiu VY, Glenn SC, Mangione CM, Sun BC. Predictors of short-term (seven-day) cardiac outcomes after emergency department visit for syncope. Am J Cardiol. 2010 Jan 1;105(1):82-6. doi: 10.1016/j.amjcard.2009.08.654. PMID 20102895
- [Background] Martin NM, Picard MH. Use and appropriateness of transthoracic echocardiography in an academic medical center: a pilot observational study. J Am Soc Echocardiogr. 2009 Jan;22(1):48-52. doi: 10.1016/j.echo.2008.10.003. Epub 2008 Nov 20. PMID 19022620
- [Background] Christopher L Moore and Joshua A Copel.